CLINICAL TRIAL: NCT04242953
Title: A Multipart Phase 1 Study to Determine Safety, Tolerability and Pharmacokinetics of SCO-120 in Healthy Male and Post-menopausal Female Subjects
Brief Title: Study to Determine Safety, Tolerability and Pharmacokinetics, of SCO-120 in Healthy Male and Post-menopausal Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SCO-120-19-18
Record Dates: First submitted 2020-01-12; First posted 2020-01-27 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteer Study

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SCO-120 (Experimental)
  Interventions: Drug: SCO-120
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: SCO-120 — Part A: single oral administration
  Part B: single oral administration in Period 1 and Period 2 (crossover design)
  Part C: multiple oral administration (14 day dosing)
  Arms: SCO-120
Drug: matching placebo — Part A: single oral administration
  Part C: multiple oral administration (14 day dosing)
  Arms: Matching Placebo

SUMMARY:
This is a Multipart Phase 1 Randomized, Double blind and Placebo controlled Study to Determine Safety, Tolerability and Pharmacokinetics, of SCO-120 in healthy male and postmenopausal female volunteers.

DETAILED DESCRIPTION:
Part A- approximately 76 (Approximately 8 sequential cohorts of 8 subjects per cohort)

Part B- Up to approximately, 32 healthy males or post-menopausal female subjects will be enrolled

Part C- Approximately 32 healthy male or postmenopausal female subjects (4 sequential cohorts of 8 subjects) will be enrolled

ELIGIBILITY:
Inclusion Criteria:

Healthy postmenopausal female volunteers will be included in the study if they meet all of the following criteria:

Part A-

1. Healthy postmenopausal female subjects, aged > 18 years, Weight over 50 kg and with a body mass index of 18.0 to 33.0 kg/m2 (inclusive) will be included in this part.
2. Did not donate 50-349 mL blood within 30 days or ≥350 mL blood within 3 months prior to IMP administration and agrees not to make blood donations, including red blood cells, plasma, platelets, or whole blood for the entire study duration.

   Part B and C-
3. Healthy male and postmenopausal female subjects, aged ≥ 18 years, with a body mass index of 18.0 to 33.0 kg/m2 (inclusive) will be included in this part.
4. Did not donate 50-499 mL blood within 30 days or ≥500 mL blood within 56 days prior to IMP administration and agrees not to make blood donations, including red blood cells, plasma, platelets, or whole blood for the entire study duration
5. Men who are able to father children must agree to use medically acceptable methods of contraception and NOT donate sperm during the study and for 90 days after the end of the study. Medically acceptable methods of contraception include using a condom with a female partner of child-bearing potential who is using oral contraceptives, hormonal patch, implant or injection, intrauterine device, or diaphragm with spermicide. Abstinence as a method of contraception is acceptable if it is in line with the preferred and usual lifestyle of the study participant.

   All parts-
6. Willing and able to give written, signed and dated informed consent (or by subject's legally acceptable representative/impartial witness when applicable) and is available for the entire study
7. Willing and able to comply with the scheduled visits, treatment plan, laboratory testing, study procedures, and restrictions (as per section 4.5), and be accessible for follow-up visits
8. Assessed as healthy based on no clinically significant abnormality identified on medical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory screening tests
9. Females who are naturally postmenopausal for at least 12 consecutive months with a follicle-stimulating hormone level of ≥ 40 mIU/mL at screening
10. Non-smokers or abstain from any tobacco usage, including smokeless tobacco, nicotine patches, etc. for entire study duration including screening period; subjects must have urine cotinine levels below those measured for smokers (< 200 ng/mL) .

Exclusion Criteria:

Subjects will be excluded from the Study if they meet any of the following criteria: (All Parts)

1. Any major surgery, as determined by the Investigator, within 4 weeks of IMP administration;
2. Blood transfusion within 4 weeks prior to IMP administration;
3. Inability to swallow oral medication;
4. Inability to undergo venipuncture and/or tolerate venous access;
5. Female on Hormone Replacement Therapy, or having been on the same in the past 6 months;
6. Active liver disease or history of liver disease (such as hepatitis) in the past 6 months which can have impact on study endpoints and/ safety of subjects as per investigator discretion;
7. Medical history of thromboembolic disorders or with risks (such as hematologic or rheumatologic disorders); recent history of thrombophlebitis;
8. Subjects with complaints of hot flashes at screening;
9. History of abnormal vaginal bleeding within 3 months prior to screening and/ or uterine malignancy
10. Positive exclusion tests: human immunodeficiency virus (HIV), hepatitis B surface antigen, or hepatitis C virus;
11. History of any relevant allergy/hypersensitivity (including known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the IMP or its excipients);
12. Received another investigational agent within 30 days (or for investigational agents with long half life a washout of 5 half-lives will be required) prior to IMP administration or intake of an investigational drug during the course of this study;
13. Intake of any prescribed medication/drugs within at least 14 days and/or over-the-counter drugs within at least 7 days (or less than 5 half-lives of the respective drug) prior to administration of the IMP;
14. Known and/ or suspected history of significant drug abuse as judged by the Investigator;
15. Positive screen for drugs of abuse at Screening visit or positive screen for alcohol or drugs of abuse on admission to the study centre prior to the first IMP administration;
16. History of alcohol abuse or excessive intake of alcohol, defined as regular weekly intake of more than 15 units of alcohol (Note: 1 unit equals 25 mL spirits, 125 mL wine, or 250 mL beer or lager) in the 12 months prior to study entry;
17. Current or recent disease of the gastrointestinal tract that may impact drug absorption and may affect the PK of the IMP, or any gastrointestinal tract surgery history that may impact drug absorption;
18. Continued use of caffeine or grapefruit juice or xanthine-containing drinks or food, e.g., coffee, tea, chocolate, red bull, or cola for 48 hours prior to dosing and till the last PK sample collection;
19. Any concomitant clinically significant disorder, like infection, diabetes etc. that would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion which can have impact on study endpoints and/ safety of subjects as per PI discretion.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Part A- Healthy postmenopausal female volunteers
  Part B & Part C- Healthy Male or postmenopausal female volunteers
Enrollment: 140 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Part A: Number of subjects with treatment-related adverse events as assessed by CTCAE version 5.0 | Day 14
  Part A: safety and tolerability assessed
Part C: Number of subjects with treatment-related adverse events as assessed by CTCAE version 5.0 | Day 35
  Part C: safety and tolerability assessed

SECONDARY OUTCOMES:
Part B: Number of subjects with treatment-related adverse events as assessed by CTCAE version 5.0 | Day 42
  Part B: safety and tolerability assessed

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - AXIS Clinicals, Dilworth, Minnesota
  - BioPharma Services USA Inc., Creve Coeur, Missouri
- BioPharma Services Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No